CLINICAL TRIAL: NCT04095130
Title: Tissue Sodium Accumulation in Patients With Psoriasis: a Pilot Study
Brief Title: Tissue Sodium in Patients With Psoriasis
Acronym: TSS1
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Heart Center (Other)
Responsible Party: Principal Investigator, Dr. Lajos Marko, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: ChariteU-ECRC-TSS1
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Psoriasis Vulgaris; Healthy
Keywords: Psoriasis; Sodium; Skin
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — human peripheral blood mononuclear cell (PBMC)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy subjects: those without a condition
  Interventions: Diagnostic Test: 23Na Magnetic resonance imaging
- Psoriasis patients: those with a condition
  Interventions: Diagnostic Test: 23Na Magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: 23Na Magnetic resonance imaging — Measurement of skin sodium content by non-invasive 23Na Magnetic resonance imaging.

SUMMARY:
Sodium can be buffered in the skin, which mechanism is altered during aging and in certain diseases such as hypertension. High salt environment can promote autoimmunity by expanding pathogenic IL-17 producing T helper (Th17) cells. Psoriasis is a relapsing and remitting inflammatory autoimmune disease affecting the skin and joints and involves proinflammatory Th17 cells. Here we tested the hypothesis if psoriatic skin has a higher sodium content in humans.

DETAILED DESCRIPTION:
The cytokine interleukin-17A (IL-17A) is a crucial player in the pathogenesis of the autoimmune disease of psoriasis. This neutrophil recruiting cytokine is produced by IL-17A producing CD4+ T cells (Th17) and gamma/delta T cells of the skin and evokes an inflammation circuit finally leading to the classical clinical picture of psoriasis with hyper- and parakeratosis, erythema, scaling and neutrophil abscess formation.

Besides genetic factors, lifestyle factors are relevant and decide if an autoimmune disease becomes manifest. It was shown previously that increased salt (sodium chloride, NaCl) concentrations boost the induction of murine and human Th17 cells. However, more - and also clinical - studies are needed to understand the correlation between salt content and IL-17A in autoimmune diseases.

This study investigates the hypothesis if skin sodium content in human psoriasis is increased in order to get further insight into the IL-17A-salt-interplay.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80
* Body mass index (BMI) 18.5- 40 kg/m2
* Glomerular filtration rate >60 ml/min/1.73m2

Exclusion Criteria:

* Diagnosed or treated hypertension and/or blood pressure above 140/90 at screening
* Palpable peripheral oedema during phyisical examination at screening
* Any type of diabetes mellitus and/or HgbA1c>6.5% at screening
* Subjects with a thyroid-stimulating hormone >4.2 mU/L at screening
* Psoriasis patients treated with systemic corticosteroids, chemotherapy agent (methothrexate) or with any kind of biologics/biosimilars
* Subjects with acute disease
* Pregnant or lactating women
* Metal or medical device implant in the body
* Tattoo on the lower extremities
* Subjects with a history of drug or alcohol abuse
* Subjects who are legal incapacitated or their circumstances do not enable the patient to fully understand the nature, significance and scope of this study.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy patients recruited locally (invitation to volunteer sent to workers of the Charié University Clinic and the Max Delbrück Center for Molecular Medicine).
  Psoriasis patients are recruited who are treated at the Department of Dermatology, Venerology and Allergology, Charité Medical Faculty, Berlin, Germany, Immanuel Krankenhaus Berlin, Medical Centre for Rheumatology and Clinical Immunology, Berlin, Germany and the Helios Clinic Berlin-Buch, Berlin, Germany.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Non-invasive sodium measurement in the skin | 4 years
  Sodium measured in the skin by 23Na-MRI is higher in psoriasis patients vs. matched healthy individuals.

CONTACTS AND LOCATIONS:
Locations (1):
- Experimental and Clinical Research Center, Clinical Research Unit, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Planned to share all IPD that underlie results in a publication.

REFERENCES:
- [Background] Kopp C, Linz P, Dahlmann A, Hammon M, Jantsch J, Muller DN, Schmieder RE, Cavallaro A, Eckardt KU, Uder M, Luft FC, Titze J. 23Na magnetic resonance imaging-determined tissue sodium in healthy subjects and hypertensive patients. Hypertension. 2013 Mar;61(3):635-40. doi: 10.1161/HYPERTENSIONAHA.111.00566. Epub 2013 Jan 21. PMID 23339169
- [Background] Kleinewietfeld M, Manzel A, Titze J, Kvakan H, Yosef N, Linker RA, Muller DN, Hafler DA. Sodium chloride drives autoimmune disease by the induction of pathogenic TH17 cells. Nature. 2013 Apr 25;496(7446):518-22. doi: 10.1038/nature11868. Epub 2013 Mar 6. PMID 23467095